CLINICAL TRIAL: NCT04055922
Title: Comparison of Solid Organ Transplant Specific and Hospital-wide Gram-Negative Antibiograms
Brief Title: Comparison of Solid Organ Transplant
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 058.PHA.2017.D
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-04

CONDITIONS: Gram-Negative Bacterial Infections; Gram-negative Bacteremia; Multidrug-Resistant Organism; Hospital-acquired Pneumonia; Healthcare-associated Pneumonia
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Solid organ transplant (SOT) recipients have increased incidence of infections with MDRO pathogens. This difference leads to a disparity in antibiograms between SOT recipients and other hospitalized patients.

DETAILED DESCRIPTION:
There is limited guidance for empiric antimicrobial therapy in this population. Local epidemiology plays a voluble role in managing infections empirically within the hospital setting. Antibiograms can serve as a critical tool in optimizing empiric antimicrobial decisions. Refining antibiogram data to specific populations such as SOT patients may allow for timelier and appropriate empiric use of antimicrobials, and improve clinical outcomes.

Time to appropriate therapy (antimicrobial testing susceptible in vitro to the pathogen identified) is of vital importance in management of serious infections. SOT may have different resistance rates at Methodist Dallas Medical Center making the applicability of the yearly hospital-wide antibiogram unknown for use in this specialized patient population. A SOT-Specific antibiogram may highlight common resistance patterns identified in pathogens seen in this patient population. Additionally, this investigation may further emphasize the importance of antimicrobial stewardship activities such as: appropriate empiric antibacterial decisions, de-escalation, and effective durations of therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

Exclusion Criteria:

* Missing data necessary to determine study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid organ transplant (SOT) recipients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Creation of a liver transplant specific antibiogram | Jan 1, 2012 - December 31, 2016
  Creation of a liver transplant specific antibiogram (cumulative susceptibility rates per bacterial organism for select antibiotics)
Creation of a kidney transplant specific antibiogram | Jan 1, 2012 - December 31, 2016
  Creation of a kidney transplant specific antibiogram (cumulative susceptibility rates per bacterial organism for select antibiotics)
Comparison of SOT | Jan 1, 2012 - December 31, 2016
  Comparison of SOT (liver and kidney) antibiograms with the hospital-wide antibiogram

SECONDARY OUTCOMES:
Creation of transplant antibiogram for subgroups | Jan 1, 2012 - December 31, 2016
  Creation of transplant antibiogram for subgroups of patients including the following: ICU patients, Kidney transplant urinary tract infections (UTI), SOT bloodstream infections (BSI)
Identification of risk factors among liver transplant recipients | Jan 1, 2012 - December 31, 2016
  Identification of risk factors among liver transplant recipients for vancomycin-resistant enterococci infections

CONTACTS AND LOCATIONS:
Overall Officials: Matt Crotty, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided